CLINICAL TRIAL: NCT04918108
Title: Inflammatory Response and Anti-inflammatory Action for Aortopathy & Arteriopathy (5A-Plan): A Multicenter Cohort Study
Brief Title: Additive Anti-inflammatory Action for Aortopathy & Arteriopathy (Multicenter Cohort Study) III
Status: Completed | Type: Observational
Sponsor: Nanjing Medical University (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other); Beijing Anzhen Hospital (Other); The Affiliated Hospital of Qingdao University (Other); First Affiliated Hospital of Shantou University Medical College (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); TEDA International Cardiovascular Hospital (Other); Xiamen Cardiovascular Hospital (Unknown); Shanghai East Hospital Tongji University (Unknown); Tianjin Chest Hospital, Tianjin Medical University (Unknown); Nanjing First Hospital, Nanjing Medical University (Other); Xiangya Hospital of Central South University (Other); The First Affiliated Hospital of Bengbu Medical University (Other)
Responsible Party: Principal Investigator, Hong Liu, Investigator of Nanjing Medical University, Nanjing Medical University
Other Study IDs: 5A Plan
Record Dates: First submitted 2021-06-03; First posted 2021-06-08 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Aortic Dissection
Keywords: Aortic Dissection; Inflammatory Response
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- inflammatory subphenotype
  Interventions: Biological: inflammatory response

INTERVENTIONS:
Biological: inflammatory response — laboratory data (leukocyte, neutrophils, monocyte, lymphocytes, platelet, fibrinogen, D-dimer, neutrophils-lymphocyte ratio, platelet-lymphocyte ratio, lymphocyte-monocyte ratio)

SUMMARY:
Anatomopathological classifications have been well identified in aortic dissection with important therapeutic implications. The authors evaluated the inflammatory response in patients with aortic dissection (AD) and assessed the presence of distinct inflammatory subphenotypes within this disease.

ELIGIBILITY:
Inclusion Criteria:

* acute type Aortic dissection;

Exclusion Criteria:

* Iatrogenic aortic dissection OR traumatic aortic dissection
* Patients with hematological diseases, infectious diseases, malignant tumors, immune system diseases, or severe liver diseases.
* Preoperative use of mechanical ventilation, blood transfusion, renal replacement therapy, extracorporeal membrane oxygenation, or intra-aortic balloon pump during the current admission.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients underwent venipuncture during primary evaluation in the Emergency Department. Venous blood samples were immediately sent to the laboratory for analysis.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
30-day mortality | 30 days after surgery
  any cause death within 30 days of surgery

SECONDARY OUTCOMES:
ICU mortality | 7 days after surgery
  any cause death within ICU

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of nanjing medical university, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu H, Zhang YY, Ding XH, Qian SC, Sun MY, Hamzah AW, Gao YN, Shao YF, Li HY, Wang K, Ni BQ, Zhang HJ; Additive Anti-inflammatory Action for Aortopathy & Arteriopathy (5A) Investigators. Proximal vs Extensive Repair in Acute Type A Aortic Dissection Surgery. Ann Thorac Surg. 2023 Aug;116(2):270-278. doi: 10.1016/j.athoracsur.2023.04.019. Epub 2023 Apr 25. PMID 37105511
- [Derived] Liu H, Qian SC, Shao YF, Li HY, Zhang HJ; 5A Investigators. Prognostic Impact of Systemic Coagulation-Inflammation Index in Acute Type A Aortic Dissection Surgery. JACC Asia. 2022 Oct 4;2(6):763-776. doi: 10.1016/j.jacasi.2022.06.007. eCollection 2022 Nov. PMID 36444319
- [Derived] Liu H, Qian SC, Han L, Dong ZQ, Shao YF, Li HY, Zhang W, Zhang HJ. Laboratory signatures differentiate the tolerance to hypothermic circulatory arrest in acute type A aortic dissection surgery. Interact Cardiovasc Thorac Surg. 2022 Nov 8;35(6):ivac267. doi: 10.1093/icvts/ivac267. PMID 36271847
- [Derived] Liu H, Qian SC, Zhang YY, Wu Y, Hong L, Yang JN, Zhong JS, Wang YQ, Wu DK, Fan GL, Chen JQ, Zhang SQ, Peng XX, Shao YF, Li HY, Zhang HJ. A Novel Inflammation-Based Risk Score Predicts Mortality in Acute Type A Aortic Dissection Surgery: The Additive Anti-inflammatory Action for Aortopathy and Arteriopathy Score. Mayo Clin Proc Innov Qual Outcomes. 2022 Sep 25;6(6):497-510. doi: 10.1016/j.mayocpiqo.2022.08.005. eCollection 2022 Dec. PMID 36185465
- [Derived] Liu H, Qian SC, Shao YF, Li HY; Additive Anti-inflammatory Action for Aortopathy & Arteriopathy (5A) Investigators Group. Anti-Inflammatory Effect of Ulinastatin on the Association Between Inflammatory Phenotypes in Acute Type A Aortic Dissection. J Inflamm Res. 2022 Jun 27;15:3709-3718. doi: 10.2147/JIR.S369703. eCollection 2022. PMID 35783246